CLINICAL TRIAL: NCT01434836
Title: Neuro-modulation of the Depressed Brain Using Working Memory Training and tDCS
Brief Title: Neuro-modulation of the Depressed Brain Using Working Memory Training and Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Presbiteriana Mackenzie (Unknown); University Ghent (Other)
Responsible Party: Principal Investigator, Andre Brunoni, Research Associate, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCS_Training
Record Dates: First submitted 2011-09-09; First posted 2011-09-15 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Depression
Keywords: Anti-depressant effects
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS and working memory training (Active Comparator)
  Interventions: Other: active tDCS and working memory training
- sham tDCS and working memory training (Placebo Comparator)
  Interventions: Other: sham tDCS and working memory training

INTERVENTIONS:
Other: active tDCS and working memory training — This group will receive 2.0 mA anodal DC stimulation over the left DLPFC and cathodal stimulation over the right DLPFC. During the stimulation, this group will be trained on working memory processes. Sessions will be scheduled daily for two consecutive weeks.
  Arms: active tDCS and working memory training
Other: sham tDCS and working memory training — This group will receive sham stimulation (e.g., identical stimulation set-up but no electric current is sent through the electrodes). Patients however receive the real working memory training, daily, for two weeks.
  Arms: sham tDCS and working memory training

SUMMARY:
The goal of this project is to train currently major depressed patients on fundamental aspects of working memory while the investigators administer transcranial Direct Current Stimulation (tDCS) over the left dorsolateral prefrontal cortex (DLPFC) during these training sessions. This working memory training would be performed using adaptive Paced Auditory Serial Addition Tasks (PASAT). The effects after two weeks of working memory training combined with tDCS or sham placebo (10 sessions) will be measured on different variables, each measured at the start and at the end of the two weeks of training. The investigators expect the greatest anti depressant results and cognitive enhancements in the group of depressed patients that received tDCS combined with working memory training.

ELIGIBILITY:
Inclusion Criteria:

* Depressive Disorder, Major (SCID)
* HDRS-24 > 21

Exclusion Criteria:

-Other axis I disorders, including Bipolar Disorder, Schizophrenia, Substance Abuse Disorders.

Any axis II disorders.

* Any serious/life-threatening axis III disorders, such as Congestive Heart Failure, Pulmonary Obstructive Chronic Disease, Active Neoplasia.
* Neurological diseases such as Stroke (and Post-Stroke Depression), Dementias and others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 4 weeks
  The primary outcome measure is the score of HDRS-24 scale after 4 weeks of treatment.

SECONDARY OUTCOMES:
Beck Depression Inventory | 4 weeks
  The outcome measure is the score of BDI scale after 4 weeks of treatment.
follow-up measure | after two weeks
  Two weeks after each participant finished his/her treatment, the investigators will contact them to verify whether treatment induces long-lasting effects. This contact will be established via email and we will ask them to fill in the same self report questionnaires as they filled in during the study protocol.
Internal Shift Task | 2 weeks
  The Internal Shift Task (IST), an emotional attention paradigm, will be administered to measure the ability to switch attention between emotional and non emotional items in working memory. After 10 sessions of tDCS in combination with the working memory training, the investigators expect a transfer effect on an increased switching ability between emotional stimuli.
Working memory task in combination with pupil dilatation | 2 weeks
  This task will be administered to measure participants' ability to manipulate emotional information in working memory: either reverse or maintain in the order of three emotion or three neutral words. The investigators hypothesize that the pupil size will be decreased when sorting negative words in working memory in depressed patients that received active tDCS over the left DLPFC in combination with attentional training.
Heart Rate Variability | 2 weeks
  This measure will be utilized to evaluate autonomic activity by recording electrocardiogram or pulse wave. High HRV has been associated with greater behavioral adaptability and plays a major role in the adaptive recovery from stress. After the treatment, the investigators expect MDD patients that received tDCS with working memory training to demonstrate increased HRV while viewing negative high arousing IAPS pictures.
Salivary Cortisol | 2 weeks
  This measure will be utilized to evaluate endocrinological response of the hypothalamic-pituitary-adrenal(HPA)axis, such as cortisol secretion. After the treatment, the investigators expect MDD patients that received tDCS with working memory training to demonstrate decreased cortisol secretion while viewing negative high arousing IAPS pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - University of São Paulo, Hospital Universitário, São Paulo, São Paulo
  - Universidade Presbiteriana Mackenzie, São Paulo, São Paulo

REFERENCES:
- [Derived] Brunoni AR, Boggio PS, De Raedt R, Bensenor IM, Lotufo PA, Namur V, Valiengo LC, Vanderhasselt MA. Cognitive control therapy and transcranial direct current stimulation for depression: a randomized, double-blinded, controlled trial. J Affect Disord. 2014 Jun;162:43-9. doi: 10.1016/j.jad.2014.03.026. Epub 2014 Mar 27. PMID 24767004